CLINICAL TRIAL: NCT06525740
Title: Methadone Versus Intrathecal Hydromorphone for Postoperative Analgesia in Patients Undergoing Surgery for Gynecologic Malignancy Via Midline Laparotomy Receiving Liposomal Bupivacaine
Brief Title: Methadone Versus Intrathecal Hydromorphone for Postoperative Pain Relief in Gynecologic Cancer Undergoing Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sean C Dowdy, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-001383; NCI-2024-06145 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-001383 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Malignant Female Reproductive System Neoplasm
MeSH Terms: interventions — Hydromorphone; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (methadone) (Experimental): Patients receive methadone IV during induction of general anesthesia for SOC surgery.
  Interventions: Drug: Methadone; Other: Questionnaire Administration
- Arm II (hydromorphone) (Experimental): Patients receive hydromorphone IT prior to induction of general anesthesia for SOC surgery.
  Interventions: Drug: Hydromorphone; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Hydromorphone — Given IT
  Other Names: (-)-Hydromorphone; Dihydromorphinone; Hydromorphon
  Arms: Arm II (hydromorphone)
Drug: Methadone — Given IV
  Arms: Arm I (methadone)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase IV trial compares methadone versus hydromorphone given in the fluid-filled space between the thin layers of tissue that cover the brain and spinal cord (intrathecal) for postoperative pain relief in patients with gynecologic cancer undergo surgery. Methadone binds to opioid receptors in the central nervous system and is a long-acting opioid pain medication. Intrathecal hydromorphone works by changing the way the brain and nervous system respond to pain and is similar to an epidural. This trial may help researchers determine if methadone works as well as intrathecal hydromorphone for pain relief after surgery in patients with gynecologic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether intravenous methadone can provide comparable analgesia to an intrathecal injection of hydromorphone.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive methadone intravenously (IV) during induction of general anesthesia for standard of care (SOC) surgery.

ARM II: Patients receive hydromorphone intrathecally (IT) prior to induction of general anesthesia for SOC surgery.

After completion of study intervention, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery with a laparotomy for gynecologic malignancy
* Planned inpatient admission greater than 24 hours

Exclusion Criteria:

* Chronic pain requiring greater than 20 morphine milligram equivalents of opioid medications as an outpatient
* Prolonged corrected QT interval (QTc) > 500ms
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) < 30 milliliters per minute (mL/min)
* Documented cirrhosis
* Preoperative platelets (PLT) < 100
* Preoperative international normalized ratio (INR) > 1.1
* Inappropriate cessation of anticoagulation medications prior to surgery
* Intolerance to hydromorphone or methadone
* Contraindication to administration of liposomal bupivacaine
* Subsequent surgeries after index surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in pain scores | Baseline, upon leaving post-anesthesia care unit (PACU), and at 4, 8, and 12 hours, up to 24 hours postoperatively
  Will be assessed per group [intravenous (IV) methadone or intrathecal (IT) hydromorphone] by patient-reported pain on a scale of 0-10 where 0=no pain and 10=worst pain imaginable.

SECONDARY OUTCOMES:
Morphine milligram equivalents | Up to 24 hours postoperatively
  Will be assessed by the number of morphine milligram equivalents utilized for the first 24 hours postoperatively.
Incidence of itching | Up to 24 hours postoperatively
  Will be assessed by the number of patients patient-reported itching on follow-up visits.
Incidence of respiratory depression | Up to 24 hours postoperatively
  Will be assessed by the number of patients who experience incidents of respiratory depression, defined breathing less frequently as a result of opioid administration.

CONTACTS AND LOCATIONS:
Overall Officials: Sean C. Dowdy, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials